CLINICAL TRIAL: NCT02099344
Title: A Prospective, Randomized Study of the Artegraft vs Propaten Vascular Grafts for Renal Failure Patients Requiring Dialysis Access
Brief Title: Artegraft Versus Propaten Dialysis Grafts
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCA-001
Record Dates: First submitted 2013-11-13; First posted 2014-03-28 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: ESRD; Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized to either
  Combination product- device/biologic Artegraft® or Gore® Propaten®.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artegraft (Active Comparator): Artegraft® vs Gore® Propaten®. Approximately 50 eligible patients with End Stage Renal Disease (ESRD) requiring hemodialysis will be randomized to receive one of these two grafts as part of their standard care.
  Interventions: Device: Artegraft
- Propaten (Active Comparator): Artegraft® vs Gore® Propaten®. Approximately 50 eligible patients with End Stage Renal Disease (ESRD) requiring hemodialysis will be randomized to receive one of these two grafts as part of their standard care.
  Interventions: Device: Propaten

INTERVENTIONS:
Device: Artegraft — Surgical placement of graft for hemodialysis access
  Arms: Artegraft
Device: Propaten — Surgical placement of graft for hemodialysis access
  Arms: Propaten

SUMMARY:
Compare Artegraft and Propaten grafts for use in dialysis access to see if one performs better than the other. How long each one lasts until a complication arises or until the graft is no longer used will be compared.

The study hypothesis is that the Artegraft, being an actual blood vessel, will work better than the manufactured Propaten graft.

DETAILED DESCRIPTION:
Approximately 50 eligible patients with End Stage Renal Disease (ESRD) requiring hemodialysis will be randomized to receive one of these two grafts as part of their standard care. Patients will be assessed at 2-3 weeks post-operatively and again at 6 and 12 months for flow characteristics, dialysis adequacy and graft associated complications such as stenosis, infection and thrombosis. Data on urea reduction ratio (URR), kinetic modeling (Kt/V), and access flow (QB) will be collected at 3, 6, 9 and 12 months via phone call to the hemodialysis center in order to evaluate patency and function.

Access complications (stenosis, thrombosis, infection) will be treated per our standard protocol. These data will be recorded and then primary, assisted primary and secondary patency rates will be calculated and the graft arms compared using life table analysis.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Candidate for hemodialysis
* Not a candidate for native AV fistula
* In need of a new AV graft in the upper arm location
* Artery and vein > 3mm.
* Medically stable and have a life expectancy of ≥ 12 months
* The patient or legal guardian understands the study and is willing to comply with the requirements.

Exclusion Criteria:

* < 18 years of age
* Current history or within 6 months of IV drug abuse
* Chronic hypotension (<100 mm systolic pressure) not responsive to treatment
* Pregnant or lactating
* Known hypercoagulable state
* Requires only a revision of an existing graft
* Receiving artery or vein is less than 3 mm in diameter at the time of implantation
* Known axillary/subclavian occlusion or stenosis that has not been treated
* Known or suspected systemic infection
* Heparin sensitivity (known HIT)
* Enrolled in another investigational study.
* Subject has more than 1 graft in target limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earl Schuman, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Propaten; Artegraft: Artegraft® vs Gore® Propaten®. Approximately 50 eligible patients with End Stage Renal Disease (ESRD) requiring hemodialysis will be randomized to receive one of these two grafts as part of their standard care.
  Artegraft: Surgical placement of graft for hemodialysis access
  Propaten: Surgical placement of graft for hemodialysis access
Period: Overall Study
Arm/Group | Propaten | Artegraft
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data not collected due to early study termination
Groups:
- Total: Total of all reporting groups
Arm/Group | Propaten | Artegraft | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 |  | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective: The Primary Objective is to Assess the Primary, Primary Assisted and Secondary Patency Rate of Each Graft
Description: The primary outcome will be determined by Kaplan-Meier life table analysis. Patency determination will be from access creation until the first occlusion of the graft.
Time Frame: 12 months
Population: Data not collected due to early study termination
Arm/Group | Propaten | Artegraft
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Examine Incidence of Complications in Patients Receiving the Artegraft Bovine Graft vs. Gore Propaten Graft
Description: Complication incidence will be collected from the time of access creation until the graft fails and is abandoned.
Time Frame: 12 months
Population: Data not collected due to early study termination
Arm/Group | Artegraft | Propaten
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: One patient enrolled, study stopped before any AE's occurred
Description: Data not collected due to early study termination
Arm/Group | Propaten | Artegraft
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No